CLINICAL TRIAL: NCT00018577
Title: The Association of Neurotoxin Exposure With Parkinson's Disease and Parkinsonism in World War II Veterans and Other Men
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: NEUD-024-99S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2004-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This program aims to investigate factors associated with development of parkinsonism or idiopathic Parkinson's Disease in an ongoing cohort of patients established in 1965 who are currently undergoing their sixth examination.

ELIGIBILITY:
This is a cohort study. Population consist of 8,006 Japanese-American men.

Min Age: 81 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 2000-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Popper, M.D.; Caroline Tanner, M.D., Ph.D.; Helen Petrovitch, M.D.; Lon White, M.D.
Locations (1):
- Honolulu Dept of Veterans Affairs, Honolulu, Hawaii, United States